CLINICAL TRIAL: NCT03297359
Title: A Multicentre Prospective Cohort Study Assessing the Use of Weight-Adjusted Low-Molecular-Weight-Heparin in Patients Over 90 kg With Acute Cancer-Associated Venous Thromboembolism
Brief Title: WAVe Study - Weight Adjusted Dalteparin for Patients Over 90 kg With Acute Cancer Associated Venous Thromboembolism
Acronym: WAVe
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WAVe-001
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cancer; Venous Thromboembolism; Obesity
Keywords: Dalteparin; Fragmin
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism; Obesity | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Weight adjusted dalteparin (Experimental): Participants will receive a daily subcutaneous injection of weight-adjusted dalteparin (See Table below) at a dose of approx. 200 IU/kg beginning on the day of enrolment and for a one month.
  91 to 95 kg: 18,000 IU daily ( or 1 prefilled syringe of 18,000 IU) 96 to 105 kg: 20,000 IU daily ( or 2 prefilled syringes of 10,000 IU) 106 to 120 kg: 22,500 IU daily ( or 2 pre-filled syringes (10,000 and 12,500 IU)) 121 to 130 kg: 25,000 IU daily ( or 2 prefilled syringes of 12,500 IU) 131 to 145 kg: 27,500 IU daily ( or 2 pre-filled syringes (12,500 and 15,000 IU)) 146 to 150 kg: 30,000 IU daily ( or 2 prefilled syringes of 15,000 IU)
  ≥ 151 kg: 33,000 IU daily ( or 2 prefilled syringes (15,000 and 18,000 IU))
  Interventions: Biological: Dalteparin

INTERVENTIONS:
Biological: Dalteparin — daily subcutaneous injection of weight-adjusted dalteparin

SUMMARY:
Cancer patients that develop blood clots are treated with low molecular weight heparin injections (LMWH). One kind of these LMWHs, dalteparin, has its dose determined based on a patient's weight using a formula of 200 international units (IU) per kilogram (kg). The current dosing of dalteparin approved by Health Canada has a maximum daily dose of 18 000 IU/day which is weight-adjusted for patients up to 90 kg. Any patient weighing more than 90 kg would take the same dosage regardless of their weight. The aim of this study is to assess the safety of using weight-adjusted dalteparin in cancer-associated venous thromboembolism patients that weigh more than 90 kg.

DETAILED DESCRIPTION:
The study is designed as a multicentre prospective cohort study with multiple Canadian sites. It will be initiated at The Ottawa Hospital prior to being offered externally. After obtaining informed consent, and confirming eligibility, participants weighing more than 90 kg with acute cancer-associated thrombosis will be treated with therapeutic weight-adjusted dalteparin (subcutaneous once daily injection, or twice daily, if the conditions of the participant do not allow once daily injection as per clinical judgement) beginning at enrolment (within 12 hours) and continuing until Day 30 visit. Subjects will receive therapeutic doses of dalteparin at a dose of approximately 200 IU/kg SC daily (up to 33,000 IU) for one month. Following this study period of 30 days (± 4 days), patients will be followed for 5 months. During the follow-up period, each patient will pursue his/her treatment as per usual standard treatment protocols provided at each institution. Treatment used and clinical outcomes will be collected at the end of the follow-up period.

The majority of Canadian Thrombosis specialists use weight adjusted dosing of dalteparin in patients weighing more than 90 kg with cancer-associated VTE. No expert recommends capping the dose of dalteparin to 18,000 IU in patients weighing over 90 kg as suggested by the product monograph. However, the risk of major bleeding episodes in patients over 90 kg receiving weight-adjusted LMWH remains unclear. The estimated rate of major bleeding episodes of patients with cancer associated VTE (Mean weight 79.1 kg) managed with therapeutic dose of dalteparin is 3.6% (95% CI: 1.9 to 6.2). We hypothesize that the rate of major bleeding events will be similar in patients (> 90 kg) with cancer-associated VTE treated with dalteparin 200 IU/kg daily (up to 33,000 IU). We plan to recruit 150 patients in this cohort study. We expect 6 major bleeding events. This would provide us with an overall bleeding event of 4% with an upper bound of the confidence interval of 8.5%). An informal survey of Canadian thrombosis expert has demonstrated that clinicians would feel reassured and continue to use weight-adjusted dalteparin in cancer patients weighing more than 90kg if the upper bound of the 95% confidence interval is less than 9% (i.e. < 3% possible absolute rate difference).

ELIGIBILITY:
Inclusion Criteria:

1. Known pathologically-confirmed cancer (other than basal-cell or squamous-cell carcinoma of the skin),
2. Confirmed symptomatic or incidental deep vein thrombosis requiring treatment, or confirmed symptomatic or incidental pulmonary embolism of a segmental or larger pulmonary artery,
3. Weight > 90 kg,
4. Age ≥18 years,
5. Hemoglobin ≥ 80 g/L,
6. Able and willing to comply with study procedures and follow-up examinations contained within the written consent form.

Exclusion Criteria:

1. Acute VTE managed with thrombectomy, insertion of an inferior vena cava filter or with the use of thrombolytic agents,
2. More than 72 hours pre-treatment with therapeutic dosage of other LMWH, direct oral anticoagulants or vitamin K antagonists prior to enrolment to manage the current VTE event (unless the participant has been treated with weight-adjusted doses of commercial dalteparin in consistency with the dosing regime outlined in the protocol up to Day 7 visit [±2 days]),
3. Contraindication to heparin therapy:

   1. history of heparin induced thrombocytopenia (HIT) as reported by patient,
   2. platelet count of less than 50 x 109/L,
   3. actively bleeding,
   4. reported history of severe uncontrolled hypertension,
   5. documented peptic ulcer within 6 weeks,
   6. reported history of severe hepatic failure,
   7. creatinine clearance of < 30 ml/min as calculated by the Cockcroft-Gault formula,
   8. heparin allergy,
   9. Other contraindication to anticoagulation.
4. An Eastern Cooperative Oncology Group (ECOG) Performance Status of 3 or 4 at the time of study enrolment,
5. Life expectancy < 1 month,
6. Women of childbearing age without proper contraceptive measures and women who are pregnant or breast feeding,
7. Participating in another interventional trial that may result in co-intervention or contamination (to be determined by sponsor),
8. Unable/unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Major bleeding episode | up to day 30
  1. Fatal bleeding, and/or,
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or,
  3. Bleeding causing a fall in hemoglobin level of ≥20 g/L, or leading to transfusion of ≥2 units of whole blood or red cells.

SECONDARY OUTCOMES:
Clinically relevant non major bleeding events | up to day 30
  As overt bleeding episodes not meeting the inclusion for major bleeding but associated with one of the following:
  1. Medical intervention,
  2. An unscheduled contact with a physician,
  3. Temporary cessation of anticoagulant treatment.
Minor bleeding events | up to day 30
  Overt bleeding not meeting the major bleeding or clinically-relevant non-major bleeding definitions
Recurrent VTE events | Up to day 180
  1. Recurrent deep vein thrombosis
  2. Recurrent Pulmonary embolism
Overall mortality | Up to day 180
  Death
Bioaccumulation of study drug | Up to day 30
  Trough anti-Xa levels measured at Day 7 and Day 30 follow-up visits will be generated for the once and twice-daily dosing regimen

CONTACTS AND LOCATIONS:
Overall Officials: Marc Carrier, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (5):
- Canada (5):
  - Alberta Health Services, Edmonton, Alberta
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hopsital, Toronto, Ontario

REFERENCES:
- [Derived] Wang TF, Yeo E, Gross PL, Seguin C, Wu C, Shivakumar S, Mallick R, Delluc A, D'Astous J, Kimpton M, Roberge G, Siegal DM, Tritschler T, Le Gal G, Carrier M. A Multicenter Prospective Cohort Study on the Use of Weight-Adjusted Dalteparin in Patients Over 90 kg With Acute Cancer-Associated Venous Thromboembolism-The WAVe Study. Am J Hematol. 2026 Jan;101(1):79-88. doi: 10.1002/ajh.70127. Epub 2025 Nov 10. PMID 41211763